CLINICAL TRIAL: NCT04059055
Title: Decreasing Unused Opioids in the Home Post Supracondylar Fracture Repair
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Conor McDonnell, Staff Anesthesiologist, The Hospital for Sick Children
Other Study IDs: 1000064960
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over the past two decades, the misuse of prescription opioids has significantly increased. A recent systematic review reported as much as 67% to 92% of opioids dispensed on discharge post-surgery go unused. This culture of overprescribing is consistently observed across surgical specialties. Less frequently observed is the potential for opioid use and misuse in children and adolescents post-surgery. The research to date in this area has been poorly performed with heterogenous data collection, analysis and reporting, as well as large loss of patients to follow-up.

The investigators' previous prospective observational deception study identified three areas of concern:

1. There is a culture of postoperative opioid over-prescribing at discharge as demonstrated by heterogenous opioid dosing and duration of treatments across practitioners for single procedures
2. This overprescribing is in excess of patients' home-requirements and results in significant quantities of leftover opioids
3. There is a culture of inappropriate storage and lack of safe disposal of prescribed opioids in the community

DETAILED DESCRIPTION:
This study focuses on addressing and minimizing pediatric surgical over-prescribing. It aims to reduce the amount of opioids prescribed by focusing prescribers and families on regular use of simple non-opioid analgesics, as well as decreasing the amount of opioids prescribed and dispensed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with supracondylar fractures undergoing surgical wire placement or pinning that return to fracture clinic at three weeks for removal of pins/wires.
* Patients discharged on the weekday.
* Families filling a prescription for opioids at Shoppers Drug Mart at SickKids Hospital.
* Parent has strong command of the English language (i.e., no interpreter required).

Exclusion Criteria:

* Patients with a history of chronic pain.
* Patient used opioid medication within the previous 6 months.
* Patients who are discharged on the weekend (as participant emails will need to be entered into redcap the day of recruitment, for data collection to commence the next morning).

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Any child (0-18 years) who has undergone a supracondylar fracture repair at The Hospital for Sick Children.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Pain medication use questionnaire | 3 days following discharge from hospital
  Recording of how many pain meds were used at home

SECONDARY OUTCOMES:
Amount of opioid returned | 3 weeks following discharge (aligns with pin/wire removal at fracture clinic)
  Recording of how much opioid was returned to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Conor Mc Donnell, Principal Investigator — Staff Anesthesiologist
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada